CLINICAL TRIAL: NCT03596489
Title: Developing a Method to Objectively Assess Sensory Nerve Fiber Sensitivity: A Pilot Study
Brief Title: Objective Assessment of Sensory Nerve Fiber Sensitivity
Status: Completed | Type: Observational
Sponsor: Julia Finkel (Other)
Responsible Party: Sponsor-Investigator, Julia Finkel, Principal Investigator, Children's National Research Institute
Organization: Children's National Research Institute (Other)
Other Study IDs: 10134
Record Dates: First submitted 2018-07-12; First posted 2018-07-24 (Actual); Last update posted 2024-07-05 (Actual); Status verified 2024-07

CONDITIONS: Nerve Pain
MeSH Terms: conditions — Neuralgia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This pilot study utilizes a unique technology to determine nerve fiber sensitivity. This will allow us to determine whether this method and device can discern changes in pain intensity and type, which is predicated on differing nerve fiber sensitivities.

ELIGIBILITY:
Inclusion Criteria:

1. The subject is 18 to 65 years of age
2. The subject is willing to have a tourniquet applied as part of the study
3. The subject is willing and able to provide written informed consent to the study participation
4. The subject is willing and able to comply with all study procedures

Exclusion Criteria:

1. Eye pathology precluding pupillometry
2. Subjects who have ongoing pain requiring medical attention
3. Subjects who are not normotensive
4. Subjects with peripheral vascular disease
5. Subjects who are morbidly obese (BMI >40)
6. Subjects with diabetes or diabetic retinopathy
7. Subjects who are or may be pregnant
8. Subjects with cardiac disease
9. Subjects with neuropathic disease states

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy Adult Volunteers will be from within the Children's National Medical Center and the surrounding community.
Sampling Method: Non-Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2018-06-27 (Actual); Primary Completion 2023-07-01 (Actual); Study Completion 2023-07-11 (Actual)

PRIMARY OUTCOMES:
Pupillary Reflex Parameters | 0,5,10,15,20,25,30,35 minutes
  The primary measurable endpoint is the change in the Area Under the Curve (AUC) of the three sensory nerve fiber types that occurs as a response to tourniquet ischemia and reperfusion. The change is calculated by the difference between measurements at various time points: baseline, tourniquet application, and tourniquet release.

CONTACTS AND LOCATIONS:
Overall Officials: Julia C Finkel, MD, Principal Investigator — Children's National Research Institute
Locations (1):
- Children's National Health System, Washington D.C., District of Columbia, United States